CLINICAL TRIAL: NCT02802163
Title: Phase I-II Study of Carfilzomib, Lenalidomide, Dexamethasone, and Panobinostat, Ca-R-Pa-Diem, as Induction Therapy for Newly Diagnosed, Untreated, Transplant-Eligible, Multiple Myeloma Patients
Brief Title: Induction Therapy for Multiple Myeloma With Carfilzomib, Lenalidomide,Dexamethasone,Panobinostat
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study drug unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18665
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
Keywords: untreated multiple myeloma; newly diagnosed myeloma; transplant eligible
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat; carfilzomib; Lenalidomide; Dexamethasone; Calcium Dobesilate; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): Combination Therapy: Panobinostat, Carfilzomib, Lenalidomide, Dexamethasone (Ca-R-Pa-Diem) . Participants will receive up to 8 cycles of the combination as induction after which will proceed with consolidation therapy with transplant as per institutional standards. After transplant, participants receive maintenance with panobinostat/lenalidomide. The maintenance dose and schedule of panobinostat will be same given during induction for 1 year. The maintenance dose of lenalidomide will be 10 mg given for 21 days of 28 days cycle until disease progression.
  Interventions: Drug: Panobinostat; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Panobinostat — Induction Phase: Panobinostat (dose escalation beginning at 10 mg) will be administered 3 times a week (TIW) by mouth every other week starting on day 1 of each cycle.
  Maintenance Phase: Panobinostat will be administered TIW by mouth every other week starting on day 1 of each cycle. The dose of panobinostat during maintenance phase will be the same dose taken during cyce 8 of induction phase.
  Other Names: LBH589; deacetylase inhibitor (DACi)
Drug: Carfilzomib — Induction Phase: Carfilzomib will be administered at 20 mg/m^2 on Cycle 1 Day 1. Beginning on Cycle 1 Day 2 the carfilzomib dose will be according to the assigned level of 27 mg/m^2 or 36 mg/m^2. Carfilzomib will be administered twice weekly IV on Days 1,2, 8,9,15, and 16.
  Other Names: Kyprolis
Drug: Lenalidomide — Induction Phase: Lenalidomide (25 mg) will be administered once-daily by mouth on Days 1-21, 25.
  Maintenance Phase: Lenalidomide (10 mg) will be administered once-daily by mouth on days 1-21.
  Other Names: Revlimid
Drug: Dexamethasone — Induction Phase: Dexamethasone (20 mg) will be administered twice weekly by mouth or by IV on Days 1,2, 8, 9, 15, and 16.
  Other Names: Decadron; corticosteroid

SUMMARY:
The purpose of this study for Phase l is to determine the maximum tolerated dose of panobinostat given in combination with carfilzomib, lenalidomide, and dexamethasone in 28-day cycles as induction (initial) therapy to participants with newly diagnosed multiple myeloma.

In Phase ll, investigators will evaluate the safety (side effects) and efficacy (effectiveness) of panobinostat in combination with carfilzomib, lenalidomide, and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years old
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Symptomatic multiple myeloma (per IMWG diagnostic criteria) and no prior treatment for multiple myeloma
* Measurable disease with at least 1 of the following assessed within 21 days prior to Cycle 1 Day 1: a.) Serum M-protein ≥ 0.5 g/d;, b.) Urine M-protein ≥ 200 mg/24 hour; c.) In potential participants without detectable serum or urine M-protein, serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal serum kappa lambda ratio.
* Must meet the following laboratory criteria within 21 days prior to Cycle 1, day 1: a.) Absolute neutrophil count (ANC) ≥ 1 x 10^9/L; b.) Hemoglobin ≥ 8 g/dl; c.) Platelet count ≥ 75,000/mm^3 unless thrombocytopenia is due to marrow infiltration by myeloma; d.) AST and ALT ≤ 2.5 x upper limit of normal (ULN); e.) Serum bilirubin ≤ 1.5 x ULN; f.) Serum Creatinine clearance ≥ 50 ml/min.
* Baseline multiple uptake gated acquisition scan (MUGA) or echocardiogram (ECHO) must demonstrate left ventricular ejection fraction (LVEF) ≥ 45%
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test within the 10 to 14 days prior to study drug administration and a negative urine pregnancy test within the 24 hours prior to the first study drug administration and males who are sexually active with FCBP must agree to use 2 highly effective concomitant methods of contraception including a male condom during the study and for 90 days following the last dose of study treatment

Exclusion Criteria:

* Prior histone deacetylase (HDAC), deacetylase (DAC), HSP90 inhibitors or valproic acid for the treatment of cancer
* Potential participants who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following: History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with principal investigator prior to enrollment); Any history of ventricular fibrillation or torsade de pointes; Bradycardia defined as HR< 50 bpm. (Patients with pacemakers are eligible if heart rate (HR) ≥ 50 bpm.); Screening ECG with a QTc > 450 msec; Right bundle branch block + left anterior hemiblock (bifascicular block); Patients with myocardial infarction or unstable angina ≤ 12 months prior to starting study drug; Other clinically significant heart disease (e.g., chronic heart failure (CHF) New York Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat
* Diarrhea > NCI common terminology criteria for adverse events (CTCAE) grade 2
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Have received prior treatment for multiple myeloma excluding dexamethasone not to exceed 160 mg total
* Have received radiation therapy to > 30% of marrow-bearing bone within < 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
* Have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test within 24 hrs of receiving the first dose of study medication.
* Males whose sexual partners are WOCBP not using effective birth control
* A prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma cell leukemia (> 2.0 × 10^9/L circulating plasma cells by standard differential)
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | Up to 8 months
  MTD of the Ca-R-Pa-Diem given in combination to newly diagnosed Multiple Myeloma patients.

SECONDARY OUTCOMES:
Stringent Complete Remission (sCR) Rate after 4 and 8 Cycles of Treatment | Up to 8 months
  Response rates by International Myeloma Working Group Uniform Response Criteria (IMWG-URC). Complete Response (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. sCR: CR plus normal free light chain (FLC) ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
Phase II: Overall Response Rate (ORR) | Up to 36 months
  Overall response rate will be the proportion of participants who achieved Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR). Response rate determined by IMWG-URC will be calculated based on the number of participants with each of response categories (sCR, CR, VGPR, PR, and progressive disease) at each treatment cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/